CLINICAL TRIAL: NCT06378957
Title: Behavioral Pharmacology of Orally Administered THC and D-limonene
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00436545
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Subjective Drug Effects; THC; D-limonene
MeSH Terms: interventions — Limonene; Dronabinol

STUDY DESIGN:
Intervention Model Description: Within-subjects design where participants are randomly assigned to dose conditions
Who Masked: Participant, Outcomes Assessor
Masking Description: place controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Oral Placebo (Placebo Comparator): Placebo (cellulose), via capsule
  Interventions: Drug: Placebo
- Oral THC 30mg (Experimental): 30mg pure THC in ethanol vehicle, via capsule
  Interventions: Drug: Delta-9-THC
- Oral THC 30mg + D-Limonene 25mg (Experimental): 30mg pure THC in ethanol vehicle, via capsule 25mg pure D-Limonene, via capsule
  Interventions: Drug: D-Limonene; Drug: Delta-9-THC
- Oral THC 30mg + D-Limonene 50mg (Experimental): 30mg pure THC in ethanol vehicle, via capsule 50mg pure D-Limonene, via capsule
  Interventions: Drug: D-Limonene; Drug: Delta-9-THC
- Oral THC 30mg + D-Limonene 100mg (Experimental): 30mg pure THC in ethanol vehicle, via capsule 100mg pure D-Limonene, via capsule
  Interventions: Drug: D-Limonene; Drug: Delta-9-THC
- Oral THC 30mg + D-Limonene 200mg (Experimental): 30mg pure THC in ethanol vehicle, via capsule 200mg pure D-Limonene, via capsule
  Interventions: Drug: D-Limonene; Drug: Delta-9-THC

INTERVENTIONS:
Drug: D-Limonene — Oral Limonene administered via capsule
  Arms: Oral THC 30mg + D-Limonene 100mg; Oral THC 30mg + D-Limonene 200mg; Oral THC 30mg + D-Limonene 25mg; Oral THC 30mg + D-Limonene 50mg
Drug: Delta-9-THC — Oral delta-9-THC in ethanol vehicle administered via capsule
  Other Names: THC
  Arms: Oral THC 30mg; Oral THC 30mg + D-Limonene 100mg; Oral THC 30mg + D-Limonene 200mg; Oral THC 30mg + D-Limonene 25mg; Oral THC 30mg + D-Limonene 50mg
Drug: Placebo — Placebo (cellulose) administered via capsule
  Arms: Oral Placebo

SUMMARY:
The current clinical trial will investigate the effects of orally administered d-limonene (limonene), delta-9-tetrahydrocannabinol (THC) and the combination in healthy adult volunteers.

DETAILED DESCRIPTION:
The current clinical trial will investigate the interaction of orally administered d-limonene (limonene) and delta-9-tetrahydrocannabinol (THC). Limonene is a flavor/fragrance component common to many plants, including cannabis. The investigators have previously demonstrated that vaporized limonene can impact the acute effects of THC. The purpose of this study is to examine whether orally administered limonene modulates the acute effects of orally co-administered THC in a manner similar to when these substances are inhaled A controlled laboratory study will be completed at Johns Hopkins evaluating placebo, THC alone, and four ascending doses of d-limonene in combination with THC. Participants will be healthy adults with experience using cannabis. A total of 6 outpatient drug administration sessions will be conducted for each evaluable participant. The investigators will recruit study volunteers until 20 participants complete the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent
* Be between the ages of 21 and 55
* Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
* Test negative for drugs of abuse other than cannabis, including breath alcohol at the screening visit and at clinic admission
* Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
* Have a body mass index (BMI) in the range of 18 to 36 kg/m2
* Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
* Have no allergies to any of the ingredients used to prepare (cellulose, THC, d-limonene).
* Report having used a high THC cannabis product in the past 3 years and having experienced anxiety after consuming cannabis at least once in lifetime.

Exclusion Criteria:

* Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine 3 month prior to the Screening Visit;
* History of or current evidence of significant medical (e.g. seizure disorder) or psychiatric illness (e.g. psychosis) judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
* Use of an over the counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
* Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
* Average use of cannabis more than 2 times per week in the prior 3 months.
* History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
* Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
* Individuals with anemia or who have donated blood in the prior 30 days

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Drug Effect as assessed by Visual Analog Scale | 8 hours after dosing
  Subjective drug effect will be measured on a 100 point visual analog scale (VAS) where 0 = no drug effect and 100 = strongest drug effect imaginable

SECONDARY OUTCOMES:
Subjective Drug Liking as assessed by Visual Analog Scale | 8 hours after dosing
  Subjective drug liking will be measured on a 100 point visual analog scale (VAS) where 0 = no drug effect and 100 = strongest drug effect imaginable
Subjective anxiety as assessed by Visual Analog Scale | 8 hours after dosing
  Subjective anxiety will be measured on a 100 point visual analog scale (VAS) where 0 = no drug effect and 100 = strongest drug effect imaginable
Subjective hunger as assessed by Visual Analog Scale | 8 hours after dosing
  Subjective hunger will be measured on a 100 point visual analog scale (VAS) where 0 = no drug effect and 100 = strongest drug effect imaginable
Subjective paranoia as assessed by Visual Analog Scale | 8 hours after dosing
  Subjective paranoia will be measured on a 100 point visual analog scale (VAS) where 0 = no drug effect and 100 = strongest drug effect imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Austin Zamarripa, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States